CLINICAL TRIAL: NCT04051112
Title: A Phase I Study Evaluating the Safety, Tolerability, Efficacy, and Pharmacokinetics of SCB-313, a Fully-Human TRAIL-Trimer Fusion Protein, for the Treatment of Malignant Ascites
Brief Title: Study With SCB-313 (Recombinant Human TRAIL-Trimer Fusion Protein) for Treatment of Malignant Ascites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Clover Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLO-SCB-313-CHN-001
Record Dates: First submitted 2019-08-04; First posted 2019-08-09 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Malignant Ascites

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCB-313 (Experimental)
  Interventions: Drug: SCB-313

INTERVENTIONS:
Drug: SCB-313 — 10mg group: Intraperitoneal injection single dose on Day 0, safety observation for 7 days, then 3 continuous doses on Day7, Day8, Day9, 21 days for 1 cycle
  Other Names: recombinant human TRAIL-Trimer fusion protein

SUMMARY:
1. The safety and tolerability of single-dose of SCB-313 will be evaluated by intraperitoneal injection;
2. The safety and tolerability of repeated-dose of SCB-313 will be evaluated by intraperitoneal injection once a day for 3 days, and the maximum tolerated dose (MTD) of SCB-313 will be determined;

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed as malignant solid tumor.
2. Malignant ascites requiring puncture drainage evaluated by investigators, defined as:

   1. if tumor cells are detectable in the ascites ,
   2. if previous surgical operation reveals extensive abdominal cavity metastasis,
   3. if there is image evidence of extensive metastasis in the abdominal cavity,
   4. if it is determined by ascites routine and ascites biochemical examination as exudate.
3. Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 3.
4. Life expectancy of at least 12 weeks.
5. Age ≥ 18 years.
6. Body weight ≥ 45 kg and body mass index (BMI) >17 kg/m2
7. Adequate hematological function, defined as: (a) Platelet count ≥100×109/L, (b) Prothrombin time and activated partial thromboplastin time ≤ 1.5 times the upper limit of normal (ULN), (c) Absolute neutrophil count ≥1.5×109/L, and (d) Hemoglobin ≥ 9 g/dL.
8. Adequate renal function, defined as serum creatinine ≤ 2.0 times ULN and creatinine clearance > 50 mL/minute.
9. Adequate liver function, defined as: (a) Aspartate aminotransferase and alanine aminotransferase ≤ 3 times ULN for patients without liver metastases, or ≤ 5 times ULN in the presence of liver metastases, and (b) Bilirubin ≤ 2.0 times ULN, unless patient has known Gilberts syndrome.
10. Albumin ≥ 2.8 g / dL (patient can use albumin to meet the standard)
11. If the serum pregnancy test of a female patient with fertility is negative within 7 days prior to the initial administration, and she is willing to use effective birth control/contraception method for contraception within 6 months after discontinuation of SCB-313.( Female patients with fertility exclude women who have undergone sterilization or menopause, which is defined as a menstrual period that lasts for one year or more without any other medical reason.) All male and female patients with reproductive potential must agree to take effective contraceptive measures during the study period and within 6 months after discontinuation of SCB-313.

    Note: Contraceptive methods considered to be effective include: complete abstinence, intrauterine devices, double barrier contraceptive methods (such as condom plus spermicide diaphragm), implanted contraceptives, hormonal contraceptives (contraceptives, implants agent, transdermal patch, hormonal vaginal device or injection for extended release), or the partner has removed the vas deferens and confirmed that it is azoospermia
12. Willing to attend follow-up visits according to study protocol.

Exclusion Criteria:

1. Loculated ascites not amenable to full drainage or benefit from abdominal treatment
2. Acute or chronic infection (such as tuberculosis) requiring antiviral or intravenous antibiotics within 2 weeks prior to enrollment.
3. Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression.
4. Residual adverse events (AEs) ≤ Grade 1 from previous treatment except alopecia.
5. Evidence or suspicion of relevant psychiatric impairment including alcohol or recreational drug abuse.
6. Myocardial infarction within 6 months prior to treatment, and/or prior diagnoses of congestive heart failure (New York Heart Association Class III or IV), unstable angina, unstable cardiac arrhythmia requiring medication, and/or long QT syndrome or QT/QTc interval >480 msec at baseline.
7. Uncontrolled hypertension defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg confirmed upon repeated measures.
8. Left ventricular ejection fraction < 50% as determined by echocardiography performed at screening
9. Hormone therapy or palliative extra abdominal radiotherapy within 1 week, prior anti-tumor therapy (chemotherapy) within 2 weeks, or other test drug within 4 weeks prior to enrollment.
10. Major surgery within 4 weeks prior to enrollment.
11. Patient with ileus within 30 days prior to screening.
12. Known portal vein obstruction (due to either prehepatic, hepatic, or posthepatic condition) which per Investigators judgement, is the primary or significant cause of ascites.
13. Positive serology test for human immunodeficiency virus type 1 and 2, or known history of other immunodeficiency disease.
14. Uncontrolled active hepatitis.
15. Scheduled participation in another clinical study involving an investigational product or device during the course of this study.
16. Previous treatment with a TRAIL-based therapy or Death Receptor (DR) 4/5 agonist therapy.
17. Known or suspected hypersensitivity to any component of the SCB 313.
18. Any further condition which, according to the investigator, may result in undue risk of the patient by participating in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-28 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
MTD | 28 days after first dosing
  MTD for single and multiple doses of SCB-313
DLT | 28 days after first dosing
  Dose Limiting Toxicity (DLT)
AE/SAE | 28 days after first dosing
  The severity of the adverse events associated with SCB-313 treatment, the incidence of serious adverse events (SAE), and the severity and incidence of adverse events (TEAE) during the DLT-observation period developed in patients, and the classification is based on the National Cancer Institute General Adverse Event Terminology

SECONDARY OUTCOMES:
Immunogenicity | Up to 28 days after first dosing
  Occurrence of binding and neutralizing anti-SCB-313 antibodies
Pharmacokinetics (Cmax) | Pre-dose(0 hour[hr]), 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr post-dose on Day 1 and Day 10
  Maximum SCB-313 concentration
Pharmacokinetics (tmax) | Pre-dose(0 hour[hr]), 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr post-dose on Day 1 and Day 10
  Time to Cmax of SCB-313
Pharmacokinetics ([AUC]0-24) | Pre-dose(0 hour[hr]), 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr post-dose on Day 1 and Day 10
  Area under SCB-313 concentration time curve from zero to 24 hours
Pharmacokinetics (AUC 0-inf) | Pre-dose(0 hour[hr]), 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr post-dose on Day 1 and Day 10
  Area under curve from time 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China